CLINICAL TRIAL: NCT03406793
Title: Randomized, Double-blind, Community-based Efficacy Trial of Various Doses of Zinc in Micronutrient Powders or Tablets in Young, Bangladeshi Children
Brief Title: Zinc-MNP Trial for Prevention of Diarrhea and Promotion of Linear Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Johns Hopkins Bloomberg School of Public Health (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1.05
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Diarrhea; Stunting
Keywords: Zinc; Multiple micronutrient powders; Diarrhea; Stunting
MeSH Terms: conditions — Diarrhea; Growth Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1. Standard MNP (Experimental)
  Interventions: Dietary Supplement: Standard MNP
- 2. High zinc, low iron MNP (Experimental)
  Interventions: Dietary Supplement: High zinc, low iron MNP
- 3. High zinc, low/no iron (Experimental)
  Interventions: Dietary Supplement: High zinc, low/no iron on alternating days
- 4. Dispersible zinc supplement (Active Comparator)
  Interventions: Dietary Supplement: Dispersible zinc supplement
- 5. Intermittent zinc supplement (Experimental)
  Interventions: Dietary Supplement: Intermittent zinc supplement
- 6. Placebo powder (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Standard MNP — Standard MNP, 15 micronutrients (Vitamin A 400 µg, vitamin D 5 µg, vitamin E 5 mg, vitamin C 30 mg, thiamine 0.5 mg, riboflavin 0.5 mg, niacin 6 mg, pyridoxine 0.5 mg, vitamin B12 0.9 mg, folate 150 µg, iron 10 mg, zinc 4.1 mg, copper 0.56 mg, selenium 17.0 µg and iodine 90 µg). Daily supplementation for 24 weeks.
  Arms: 1. Standard MNP
Dietary Supplement: High zinc, low iron MNP — Same as group 1, except with 10 mg zinc instead of 4.1 mg and 6 mg iron instead of 10 mg. Daily supplementation for 24 weeks.
  Arms: 2. High zinc, low iron MNP
Dietary Supplement: High zinc, low/no iron on alternating days — Same as study group 1, except with 10 mg zinc instead of 4.1 mg, and 6 mg iron and no iron on alternating days instead of 10 mg. Daily supplementation for 24 weeks.
  Arms: 3. High zinc, low/no iron
Dietary Supplement: Dispersible zinc supplement — 10 mg zinc in a dispersible tablet. Daily supplementation for 24 weeks.
  Arms: 4. Dispersible zinc supplement
Dietary Supplement: Intermittent zinc supplement — 10 mg zinc in a dispersible tablet. Daily supplementation for 14 days at baseline and 3 months, placebo tablet on all other days.
  Arms: 5. Intermittent zinc supplement
Dietary Supplement: Placebo powder — Daily provision of a placebo powder for 24 weeks.
  Arms: 6. Placebo powder

SUMMARY:
This is a randomized, double-blind, community-based efficacy trial of different doses, forms, and frequencies of zinc supplementation for the prevention of diarrhea and promotion of linear growth among children 9-11 months of age in Dhaka, Bangladesh.

DETAILED DESCRIPTION:
Zinc is essential to support growth in young children especially for tissues undergoing rapid cellular differentiation and turnover, such as those in the immune system and gastrointestinal tract. Therapeutic zinc supplementation has been initiated in low-income countries as part of diarrhea treatment programs to support these needs for young children but, the effects of preventive supplemental zinc as a tablet or as a multiple micronutrient powder (MNP) on child growth and diarrheal disease are mixed and pose programmatic uncertainties. Thus, a randomized, double-blind community-based efficacy trial of five different doses, forms, and frequencies of preventive zinc supplementation vs. a placebo was designed for a study in children aged 9-11 months in an urban community in Dhaka, Bangladesh. The primary outcomes of this 24-week study are incidence of diarrheal disease and linear growth. Study workers will conduct in-home morbidity checks twice weekly; anthropometry will be measured at baseline, 12 weeks and 24 weeks. Serum zinc and other related biomarkers will be measured in a subsample along with an estimate of the exchangeable zinc pool size using stable isotope techniques in a subgroup. Therapeutic zinc will be provided as part of diarrhea treatment, in accordance with Bangladesh's national policy. Therefore, the proposed study will determine the additional benefit of a preventive zinc supplementation intervention.

ELIGIBILITY:
Inclusion Criteria:

* 9-11 months of age
* Weight-for-length Z score >= -3 according to the 2006 World Health Organization Growth Standards
* Hemoglobin concentration > = 7.0 g/dL

Exclusion Criteria:

* Presence of severe acute malnutrition, defined as a WLZ <-3 and/or the presence of bipedal edema and/or mid-upper arm circumference <115 mm;
* Presence of severe anemia, defined as a hemoglobin concentration < 7.0 g/dL
* Congenital anomalies (e.g. cardiac defects, cleft lip or palate) or any other conditions that interfere with feeding;
* Chromosomal anomalies and other organic problems (e.g. jaundice, tuberculosis)
* Currently consuming MNPs with no intention of stopping

Ages: 9 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2886 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrhea | Incidence over the 24-week follow-up period
  Incidence of diarrhea is defined as the number of diarrheal episodes per person-weeks of follow-up
Change in length-for-age Z score | Measured at enrollment and the end of the 24-week follow-up period
  Change in length-for-age Z score from enrollment to the end of the 24-week follow-up period

SECONDARY OUTCOMES:
Change in stunting prevalence | Measured at enrollment and the end of the 24-week follow-up period
  Change in the prevalence of stunting (LAZ <-2) in the study population over the 24-week follow-up period
Change in wasting prevalence | Measured at enrollment and at the end of the 24-week follow-up period
  Change in the prevalence of wasting (WLZ <-2) in the study population over the 24-week follow-up period
Incidence of dysentery | Measured twice weekly for 24 weeks
  Dysentery is defined as any diarrheal episode in which the loose or watery stools contain visible red blood
Incidence of diarrhea with dehydration | Measured twice weekly for 24 weeks
  Incidence of diarrhea with dehydration over the 24-week follow-up period
Incidence of hospitalizations | Assessed twice weekly for 24 weeks
  Hospitalization is defined as an overnight stay in the hospital due to illness
Change in mean serum zinc concentration | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants in all 6 intervention groups
  Change in mean serum zinc concentration among children in the biochemistry sub-group over the 24-week follow-up period
Change in the prevalence of zinc deficiency | Measured at enrollment and at the end of the 24-week follow-up period in subgroup of participants in all 6 intervention groups
  Change in the prevalence of zinc deficiency (serum zinc concentration <9.9 umol/L) in the biochemistry subgroup from baseline to the end of the 24-week follow-up period
Change in the exchangeable zinc pool size | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  Change in the exchangeable zinc pool size from enrollment to the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP group, dispersible zinc supplement group, and placebo group
Change in ferritin concentrations | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants in all 6 intervention groups
  Change in mean concentrations of ferritin from enrollment to the end of the 24-week follow-up period among participants in the biochemistry subgroup.
Change in concentrations of soluble transferrin receptor | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants in all 6 intervention groups
  Change in mean concentrations of soluble transferrin receptor from enrollment to the end of the 24-week follow-up period among participants in the biochemistry subgroup.
Change in gut microbiota | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  Change in the composition of gut microbiota from enrollment to the end of the 24-week follow-up period among a subgroup of participants randomized to the high zinc, low-iron; dispersible zinc supplement; and placebo powder groups.
Change in amino acid metabolites associated with gut permeability | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  To compare the change in amino acid metabolites associated with gut permeability from enrollment to the end of the 24-week follow-up period among a subgroup of participants randomized to the high zinc, low-iron MNP; dispersible zinc supplement; and placebo groups.
Change in lipid metabolites associated with gut permeability | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  To compare the change in lipid metabolites associated with gut permeability from enrollment to the end of the 24-week follow-up period among a subgroup of participants randomized to the high zinc, low-iron MNP; dispersible zinc supplement; and placebo groups.
Change in genome wide gene expression by RNA-sequencing | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  To compare the change in genome wide gene expression, measured with RNA-sequencing, from enrollment to the end of the 24-week follow-up period among a subgroup of participants randomized to the high zinc, low-iron MNP; dispersible zinc supplement; and placebo groups.
Change in specific gene expression by quantitative Polymerase Chain Reaction | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  To compare the change in specific gene expression, measured by quantitative Polymerase Chain Reaction, from enrollment to the end of the 24-week follow-up period among a subgroup of participants randomized to the high zinc, low-iron MNP; dispersible zinc supplement; and placebo groups.
Change in cellular immune function by leukocyte profiles | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  To compare the change in cellular immune function by leukocyte profiles, from enrollment to the end of the 24-week follow-up period among a subgroup of participants randomized to the high zinc, low-iron MNP; dispersible zinc supplement; and placebo groups.
Change in serum cytokines | Measured at enrollment and at the end of the 24-week follow-up period in a subgroup of participants randomized to the high zinc, low-iron MNP, dispersible zinc supplement, and placebo groups.
  To compare the change in serum cytokines, measured by Luminex analysis, from enrollment to the end of the 24-week follow-up period among a subgroup of participants randomized to the high zinc, low-iron MNP; dispersible zinc supplement; and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Black, MD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Islam MM, Black RE, Krebs NF, Westcott J, Long J, Islam KM, Peerson JM, Sthity RA, Khandaker AM, Hasan M, El Arifeen S, Ahmed T, King JC, McDonald CM. Different Doses, Forms, and Frequencies of Zinc Supplementation for the Prevention of Diarrhea and Promotion of Linear Growth among Young Bangladeshi Children: A Six-Arm, Randomized, Community-Based Efficacy Trial. J Nutr. 2022 May 5;152(5):1306-1315. doi: 10.1093/jn/nxab439. PMID 35015856